CLINICAL TRIAL: NCT03507231
Title: Non-integrated Costs Increase Effectiveness of Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: Rutgers University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P30AG0345462017
Record Dates: First submitted 2018-01-24; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Control - No Incentive for Flu Vaccine; Direct Incentive; Indirect Incentive
Keywords: incentives; field study; vaccination
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants will receive an E-mail Message encouraging them to get vaccinated, and asking them to indicate if they intend to do so and to complete a brief questionnaire after vaccination.
  Interventions: Behavioral: Email Message
- Direct Incentive (Experimental): Participants will receive an E-mail Message encouraging them to get vaccinated, and asking them to indicate if they intend to do so and to complete a brief questionnaire after vaccination. They are offered an Incentive for Vaccination ($5 Amazon Gift Card).
  Interventions: Behavioral: Email Message; Behavioral: Incentive for Vaccination
- Indirect Incentive (Experimental): Participants will receive an E-mail Message encouraging them to get vaccinated, and asking them to indicate if they intend to do so and to complete a brief questionnaire after vaccination. They are offered an Incentive for completing a short survey ($5 Amazon Gift Card).
  Interventions: Behavioral: Email Message; Behavioral: Incentive for completing a short survey

INTERVENTIONS:
Behavioral: Email Message — Participants will randomly receive an e-mail message about the availability of free flu vaccines.
Behavioral: Incentive for Vaccination — $5 gift card offered for vaccination
  Arms: Direct Incentive
Behavioral: Incentive for completing a short survey — $5 gift card offered for completing s short survey after one gets vaccinated
  Arms: Indirect Incentive

SUMMARY:
The investigators will test the hypothesis that the control (no incentive) condition will have the lowest vaccination rate, the main task condition will have a significantly higher vaccination rate while the indirect condition will have the highest vaccination rate.

Participants will be randomly assigned to one of the three message conditions and their vaccination records obtained from the university Occupational Health Department.

DETAILED DESCRIPTION:
The investigators will send e-mails to a complete mailing list of faculty and staff at a university. Each recipient will be randomly assigned to one of three conditions: control, main task incentive or indirect incentive. Our main dependent variable will be whether or not participants decide to get vaccinated. The investigators will obtain their actual vaccination records from the university Occupational Health Department.

Within the e-mail message, participants will indicate whether or not they intend to get vaccinated. Intention serves as an indirect dependent outcome. Upon clicking to indicate their intention, participants are redirected to a page which gives further instructions on how to proceed.

Participants who vaccinate will be asked to complete a brief follow-up questionnaire to evaluate their experience with vaccination and (for those offered and incentive) to provide contact information to receive their payment.

ELIGIBILITY:
Inclusion Criteria:

* Must be faculty or staff at Rutgers University.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12531 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Number of people vaccinated | Up to 5 months
  Measure the number of people who got vaccinated in the Fall 2017 semester at a large state university. We will collect vaccination records from the university Occupational Health Department

SECONDARY OUTCOMES:
Intention to get vaccinated | Up to 5 months
  Participants will receive an e-mail with our main treatment manipulations. In each e-mail they will be able to indicate whether or not they want to get vaccinated. We will use this measure as a second dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: George Loewenstein, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (condition, vaccination status) will be shared on a site such as Open Science Framework
Supporting Information: Analytic Code
Time Frame: 12/31/2019, indefinitely
Access Criteria: open access
URL: https://osf.io/

REFERENCES:
- [Background] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Result] Chapman GB, Li M, Colby H, Yoon H. Opting in vs opting out of influenza vaccination. JAMA. 2010 Jul 7;304(1):43-4. doi: 10.1001/jama.2010.892. No abstract available. PMID 20606147